CLINICAL TRIAL: NCT06416436
Title: Immunotherapy in Combination With Ablative Radiosurgery to Ultra-high DoSes (ICARUS): A Phase I Dose-escalation Radiosurgery Study in Metastatic Cancers
Brief Title: Dose-escalation Study of Ultra-high Dose Ablative Radiosurgery With Immunotherapy for Bulky Metastatic Cancer Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Impasse during contract negotitations
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-ICARUS
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
Keywords: Stereotactic Ablative Radiotherapy; SBRT; Atezolizumab; Tecentriq; Metastatic; Phase I
MeSH Terms: conditions — Neoplasm Metastasis | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Traditional 3+3 model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SBRT with concurrent and adjuvant atezolizumab immunotherapy (Experimental)
  Interventions: Drug: Atezolizumab; Radiation: Stereotactic Ablative Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose of 1680 mg IV route every 4 weeks (1680 mg on Day 1 of each 28-day cycle), which is an approved dosage for atezolizumab, as outlined in the prescribing information.
Radiation: Stereotactic Ablative Radiotherapy (SBRT) — Ultra-High Doses of Ablative Radiosurgery
  SBRT is delivered to metastases over 3-5 fractions within 1-2 weeks

SUMMARY:
The purpose of this study is to determine whether cytoreduction of bulky metastatic disease using ultra high dose SBRT in combination with immunotherapy is tolerable and feasible In patients who have exhausted SoC treatment options.

DETAILED DESCRIPTION:
Patients that provide informed consent will undergo a 30-day screening period to determine eligibility for the trial. If eligible, patients will begin treatment on SBRT (delivered to metastases over 3-5 fractions within 1-2 weeks) with concurrent and adjuvant atezolizumab (1680 mg on Day 1 of each 28-day cycle) immunotherapy regimen for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to understand this study, and participant willingness to sign a written informed consent
* Males and females age ≥ 18 years
* Measurable disease by RECIST 1.1 Participants must have at least two radiographically identifiable lesions measurable by RECIST v1.1 criteria and one of those lesions must be ≥65 cc. NOTE: 'cc' equals (width x length x height)/2 to provide rough approximation. For example, a 5.1 x 5.1 x 5.1 cm tumor would be 66.3 cc and appropriate for trial enrollment
* Participants must have washout period of 5 elimination half-lives or 28 days (whichever is longer) from time of last systemic therapy to start of study treatment
* Women of childbearing potential must have a negative serum pregnancy test at time of enrollment (at screening and up to 48 hours prior to start of radio- or immuno- therapy)
* Participants with biopsy and radiographically confirmed metastatic cancer (i.e., Lung, head and neck, ovarian, colorectal, sarcoma)
* At least 1st line (1L) systemic therapy or immunotherapy must have failed for participants and standard of care therapy options must also be exhausted. Standard of care options that have been discontinued for reasons other than disease progression are eligible. NOTE: Participants who are off systemic therapy who are being monitored with surveillance imaging, who then develop disease progression and are without standard of care therapy options are eligible for enrollment.
* At least one lesion (and up to a maximum of four lesions) must be ≥65 cc (calculated using tumor length x width x height to closest approximation)
* Prior RT is permitted if the lesion to be treated and surrounding region (no appreciable dosimetric overlap, assessed on case-by-case basis as needed) with ultra-high dose SBRT was not previously treated
* Participants with CNS metastatic disease will be allowed on protocol if all lesions are managed prior to starting extra-CNS ablative therapy
* Availability of a representative (FFPE) tumor specimen from metastatic diagnosis of cancer done prior to any study intervention for exploratory study-related biomarker research
* Adequate organ function, defined as the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  1. Leukocytes ≥ 3K/µL
  2. Lymphocyte count ≥ 0.5 x 10^9/L (500/µL)
  3. Absolute Neutrophil Count ≥1.5K/µL without granulocyte colony-stimulating factor support. NOTE: Participants with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 if in the opinion of treating physician the trial treatment does not pose excessive risk of infection to the participant
  4. Platelets ≥100K/μL) without transfusion
  5. Hemoglobin ≥ 9 g/dL
  6. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) [calculated using the Cockcroft-Gault formula]
  7. Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN. Participants with known Gilbert disease: serum bilirubin ≤ 3 x ULN
  8. Serum albumin ≥ 35 g/L (3.5 g/dL)
  9. Aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
  10. For participants not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN
  11. For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
  12. Negative HIV test at screening, with the following exception: Participants with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/µL, and have an undetectable viral load. *** NOTE: A participant may be eligible if test is positive and will be left to the investigator to determine appropriateness for trial enrollment if medically stable and without signs of active, uncontrolled disease. Prior to formal enrollment, please contact protocol study PI to review.
  13. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test must be performed for participants who have a positive HCV antibody test.*** NOTE: A participant may be eligible if test is positive and will be left to the investigator to determine appropriateness for trial enrollment if medically stable and without signs of active, uncontrolled disease. Prior to formal enrollment, please contact protocol study PI to review.
  14. Negative hepatitis B surface antigen (HbsAg) test at screening. Negative total hepatitis B core antibody (HbcAb) test at screening, or positive total HbcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for participants who have a negative HbsAg test and a positive total HbcAb test. *** NOTE: A participant may be eligible if test is positive and will be left to the investigator to determine appropriateness for trial enrollment if medically stable and without signs of active, uncontrolled disease. Prior to formal enrollment, please contact protocol study PI to review.
  15. Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section and below for the duration of study participation and for 180 DAYS/6 MONTHS following completion of therapy. Men must refrain from donating sperm during this same period.

      1. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a woman with a tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
      2. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
      3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

Exclusion Criteria:

* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Is pregnant or breastfeeding
* Female of childbearing potential planning to become pregnant while receiving study treatment or for less than 180 DAYS/6 MONTHS after the last dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result at time of enrollment (at screening and up to 48 hours prior to start of radio- or immuno- therapy).
* Male of childbearing potential planning to father a child or donate sperm while receiving study treatment or for less than 180 DAYS / 6 MONTHS after the last dose of study treatment
* Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment
* COVID-19: Participants with active COVID-19 symptoms and/or hospitalized for severe or critical COVID-19 symptoms
* Participants with uncontrolled concurrent illness or infection (i.e., active pneumonia or infection)
* Participants with only bone metastatic disease
* Immunosuppressive disorders (i.e., solid organ transplant recipient, allogeneic stem cell transplant) (please refer Appendix D for full list)
* Participants who are enrolled in hospice or felt to have less than 6 months life expectation
* Uncontrolled or untreated CNS metastases

  1. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
  2. Asymptomatic participants with treated CNS lesions are eligible, provided that all of the following criteria are met:

     1. Measurable disease, per RECIST v1.1, must be present outside the CNS
     2. The participant has no history of intracranial hemorrhage or spinal cord hemorrhage
     3. The participant has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
     4. The participant has no ongoing requirement for corticosteroids as therapy for CNS disease
     5. If the participant is receiving anti-convulsant therapy, the dose is considered stable
* History of leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). • Participants with indwelling catheters (e.g., PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN
* Uncontrolled tumor-related pain. Participants requiring pain medication must be on a stable regimen at study entry.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, scleroderma, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  1. Participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study
  2. Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  3. Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

     1. Rash must cover < 10% of body surface area
     2. Disease is well controlled at baseline and requires only low-potency topical corticosteroids
     3. There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
  4. See also Appendix D for list of autoimmune diseases and immune deficiencies
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact participant safety
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Participants receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with checkpoint blockade therapy
* History of prior immunotherapy induced pneumonitis and/or peritonitis that is Grade ≥3 is not permitted (instance of Grade 1 or 2 that have fully recovered and tolerated subsequent immunotherapy is permitted)
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  1. Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study
  2. Participants who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the atezolizumab formulation
* Has a known allergic reaction to any excipient contained in the study drug formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ultra-high dose Stereotactic Ablative Radiotherapy (SBRT) for 3 different body sites | 1 Month
  Maximum tolerated dose of ultra-high dose SBRT for 3 different body sites (i.e., peripheral lung, mediastinum-central lung, and abdomen-pelvis)

SECONDARY OUTCOMES:
Evaluate the number of participants receiving ultra-high dose ablative radiosurgery with immunotherapy who develop treatment-related adverse events as assessed by CTCAE v4.0 | Enrollment to 1 month after end of SBRT treatment (approximately 2 months)
  To assess the safety of ultra-high dose SBRT with concurrent and adjuvant atezolizumab in participants with cancer who have exhausted standard of care treatment options
Overall tumor response rate to ultra-high dose SBRT for 3 different body sites | Pre-treatment to 3 and 6 months after SBRT (approximately 7 months)
  To assess the overall tumor response rate of participants receiving ultra-high dose SBRT with concurrent and adjuvant atezolizumab
Progression-Free Survival of participants receiving ultra-high dose Stereotactic Ablative Radiotherapy (SBRT) with concurrent and adjuvant atezolizumab | Up to 2 years
  To assess the progression-free survival of participants receiving ultra-high dose SBRT with concurrent and adjuvant atezolizumab in participants with cancer who have exhausted standard of care treatment options.
Overall Survival of participants receiving ultra-high dose Stereotactic Ablative Radiotherapy (SBRT) with concurrent and adjuvant atezolizumab | Up to 2 years
  To assess the overall survival of participants receiving ultra-high dose SBRT with concurrent and adjuvant atezolizumab in participants with cancer who have exhausted standard of care treatment options

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Gan, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Ganesh K, Massague J. Targeting metastatic cancer. Nat Med. 2021 Jan;27(1):34-44. doi: 10.1038/s41591-020-01195-4. Epub 2021 Jan 13. PMID 33442008
- [Background] Corkum MT, Rodrigues GB. Patient selection for thoracic radiotherapy in extensive-stage small-cell lung cancer. Lung Cancer Manag. 2017 Nov;6(2):47-53. doi: 10.2217/lmt-2017-0006. Epub 2017 Nov 17. PMID 30643570
- [Background] Lutz ST, Jones J, Chow E. Role of radiation therapy in palliative care of the patient with cancer. J Clin Oncol. 2014 Sep 10;32(26):2913-9. doi: 10.1200/JCO.2014.55.1143. Epub 2014 Aug 11. PMID 25113773
- [Background] Rodrigues G, Videtic GM, Sur R, Bezjak A, Bradley J, Hahn CA, Langer C, Miller KL, Moeller BJ, Rosenzweig K, Movsas B. Palliative thoracic radiotherapy in lung cancer: An American Society for Radiation Oncology evidence-based clinical practice guideline. Pract Radiat Oncol. 2011 Apr-Jun;1(2):60-71. doi: 10.1016/j.prro.2011.01.005. Epub 2011 Apr 8. PMID 25740118
- [Background] 8 Gy single fraction radiotherapy for the treatment of metastatic skeletal pain: randomised comparison with a multifraction schedule over 12 months of patient follow-up. Bone Pain Trial Working Party. Radiother Oncol. 1999 Aug;52(2):111-21. PMID 10577696
- [Background] Waldman AD, Fritz JM, Lenardo MJ. A guide to cancer immunotherapy: from T cell basic science to clinical practice. Nat Rev Immunol. 2020 Nov;20(11):651-668. doi: 10.1038/s41577-020-0306-5. Epub 2020 May 20. PMID 32433532
- [Background] Hendry S, Salgado R, Gevaert T, Russell PA, John T, Thapa B, Christie M, van de Vijver K, Estrada MV, Gonzalez-Ericsson PI, Sanders M, Solomon B, Solinas C, Van den Eynden GGGM, Allory Y, Preusser M, Hainfellner J, Pruneri G, Vingiani A, Demaria S, Symmans F, Nuciforo P, Comerma L, Thompson EA, Lakhani S, Kim SR, Schnitt S, Colpaert C, Sotiriou C, Scherer SJ, Ignatiadis M, Badve S, Pierce RH, Viale G, Sirtaine N, Penault-Llorca F, Sugie T, Fineberg S, Paik S, Srinivasan A, Richardson A, Wang Y, Chmielik E, Brock J, Johnson DB, Balko J, Wienert S, Bossuyt V, Michiels S, Ternes N, Burchardi N, Luen SJ, Savas P, Klauschen F, Watson PH, Nelson BH, Criscitiello C, O'Toole S, Larsimont D, de Wind R, Curigliano G, Andre F, Lacroix-Triki M, van de Vijver M, Rojo F, Floris G, Bedri S, Sparano J, Rimm D, Nielsen T, Kos Z, Hewitt S, Singh B, Farshid G, Loibl S, Allison KH, Tung N, Adams S, Willard-Gallo K, Horlings HM, Gandhi L, Moreira A, Hirsch F, Dieci MV, Urbanowicz M, Brcic I, Korski K, Gaire F, Koeppen H, Lo A, Giltnane J, Rebelatto MC, Steele KE, Zha J, Emancipator K, Juco JW, Denkert C, Reis-Filho J, Loi S, Fox SB. Assessing Tumor-infiltrating Lymphocytes in Solid Tumors: A Practical Review for Pathologists and Proposal for a Standardized Method From the International Immunooncology Biomarkers Working Group: Part 1: Assessing the Host Immune Response, TILs in Invasive Breast Carcinoma and Ductal Carcinoma In Situ, Metastatic Tumor Deposits and Areas for Further Research. Adv Anat Pathol. 2017 Sep;24(5):235-251. doi: 10.1097/PAP.0000000000000162. PMID 28777142
- [Background] Miyashita M, Sasano H, Tamaki K, Hirakawa H, Takahashi Y, Nakagawa S, Watanabe G, Tada H, Suzuki A, Ohuchi N, Ishida T. Prognostic significance of tumor-infiltrating CD8+ and FOXP3+ lymphocytes in residual tumors and alterations in these parameters after neoadjuvant chemotherapy in triple-negative breast cancer: a retrospective multicenter study. Breast Cancer Res. 2015 Sep 4;17(1):124. doi: 10.1186/s13058-015-0632-x. PMID 26341640
- [Background] Yang C, Jin J, Yang Y, Sun H, Wu L, Shen M, Hong X, Li W, Lu L, Cao D, Wang X, Sun J, Ye Y, Su B, Deng L. Androgen receptor-mediated CD8+ T cell stemness programs drive sex differences in antitumor immunity. Immunity. 2022 Jul 12;55(7):1268-1283.e9. doi: 10.1016/j.immuni.2022.05.012. Epub 2022 Jun 13. PMID 35700739
- [Background] Ying L, Yan F, Meng Q, Yu L, Yuan X, Gantier MP, Williams BRG, Chan DW, Shi L, Tu Y, Ni P, Wang X, Chen W, Zang X, Xu D, Hu Y. PD-L1 expression is a prognostic factor in subgroups of gastric cancer patients stratified according to their levels of CD8 and FOXP3 immune markers. Oncoimmunology. 2018 Feb 20;7(6):e1433520. doi: 10.1080/2162402X.2018.1433520. eCollection 2018. PMID 29872566
- [Background] Ribas A, Wolchok JD. Cancer immunotherapy using checkpoint blockade. Science. 2018 Mar 23;359(6382):1350-1355. doi: 10.1126/science.aar4060. Epub 2018 Mar 22. PMID 29567705
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Baumeister SH, Freeman GJ, Dranoff G, Sharpe AH. Coinhibitory Pathways in Immunotherapy for Cancer. Annu Rev Immunol. 2016 May 20;34:539-73. doi: 10.1146/annurev-immunol-032414-112049. Epub 2016 Feb 25. PMID 26927206
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Garcia-Diaz A, Shin DS, Moreno BH, Saco J, Escuin-Ordinas H, Rodriguez GA, Zaretsky JM, Sun L, Hugo W, Wang X, Parisi G, Saus CP, Torrejon DY, Graeber TG, Comin-Anduix B, Hu-Lieskovan S, Damoiseaux R, Lo RS, Ribas A. Interferon Receptor Signaling Pathways Regulating PD-L1 and PD-L2 Expression. Cell Rep. 2017 May 9;19(6):1189-1201. doi: 10.1016/j.celrep.2017.04.031. PMID 28494868
- [Background] Nimmagadda S. Quantifying PD-L1 Expression to Monitor Immune Checkpoint Therapy: Opportunities and Challenges. Cancers (Basel). 2020 Oct 29;12(11):3173. doi: 10.3390/cancers12113173. PMID 33137949
- [Background] Bae SH, Kim MS, Cho CK, Kang JK, Kang HJ, Kim YH, Shin US, Moon SM, Lee DH. High dose stereotactic body radiotherapy using three fractions for colorectal oligometastases. J Surg Oncol. 2012 Aug 1;106(2):138-43. doi: 10.1002/jso.23058. Epub 2012 Feb 1. PMID 22297789
- [Background] Marzo AD, Casale M, Trippa F, Anselmo P, Arcidiacono F, Draghini L, Terenzi S, Maranzano E. Stereotactic Body Radiotherapy in Contralateral Kidney Oligometastasis From Renal Cell Carcinoma in a Nephrectomized Patient. Ochsner J. 2021 Fall;21(3):296-300. doi: 10.31486/toj.20.0080. PMID 34566513
- [Background] Ogawa Y, Shibamoto Y, Hashizume C, Kondo T, Iwata H, Tomita N, Ogino H. Repeat stereotactic body radiotherapy (SBRT) for local recurrence of non-small cell lung cancer and lung metastasis after first SBRT. Radiat Oncol. 2018 Jul 28;13(1):136. doi: 10.1186/s13014-018-1080-4. PMID 30055636
- [Background] Oura S, Mori M, Makimoto S. A Case of Solitary Lung Metastasis of Breast Cancer Successfully Treated with Stereotactic Body Radiotherapy after Chemotherapy. Case Rep Oncol. 2020 Apr 9;13(1):398-402. doi: 10.1159/000506733. eCollection 2020 Jan-Apr. PMID 32355496
- [Background] Weykamp F, Konig L, Seidensaal K, Forster T, Hoegen P, Akbaba S, Mende S, Welte SE, Deutsch TM, Schneeweiss A, Debus J, Horner-Rieber J. Extracranial Stereotactic Body Radiotherapy in Oligometastatic or Oligoprogressive Breast Cancer. Front Oncol. 2020 Jun 26;10:987. doi: 10.3389/fonc.2020.00987. eCollection 2020. PMID 32676455
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Weichselbaum RR. The 46th David A. Karnofsky Memorial Award Lecture: Oligometastasis-From Conception to Treatment. J Clin Oncol. 2018 Nov 10;36(32):3240-3250. doi: 10.1200/JCO.18.00847. Epub 2018 Sep 27. PMID 30260759
- [Background] Hughes KS, Simon R, Songhorabodi S, Adson MA, Ilstrup DM, Fortner JG, Maclean BJ, Foster JH, Daly JM, Fitzherbert D, et al. Resection of the liver for colorectal carcinoma metastases: a multi-institutional study of patterns of recurrence. Surgery. 1986 Aug;100(2):278-84. PMID 3526605
- [Background] Nordlinger B, Guiguet M, Vaillant JC, Balladur P, Boudjema K, Bachellier P, Jaeck D. Surgical resection of colorectal carcinoma metastases to the liver. A prognostic scoring system to improve case selection, based on 1568 patients. Association Francaise de Chirurgie. Cancer. 1996 Apr 1;77(7):1254-62. PMID 8608500
- [Background] Fong Y, Fortner J, Sun RL, Brennan MF, Blumgart LH. Clinical score for predicting recurrence after hepatic resection for metastatic colorectal cancer: analysis of 1001 consecutive cases. Ann Surg. 1999 Sep;230(3):309-18; discussion 318-21. doi: 10.1097/00000658-199909000-00004. PMID 10493478
- [Background] Pawlik TM, Scoggins CR, Zorzi D, Abdalla EK, Andres A, Eng C, Curley SA, Loyer EM, Muratore A, Mentha G, Capussotti L, Vauthey JN. Effect of surgical margin status on survival and site of recurrence after hepatic resection for colorectal metastases. Ann Surg. 2005 May;241(5):715-22, discussion 722-4. doi: 10.1097/01.sla.0000160703.75808.7d. PMID 15849507
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Griffioen G, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Bauman GS, Warner A, Senan S. Stereotactic ablative radiotherapy versus standard of care palliative treatment in patients with oligometastatic cancers (SABR-COMET): a randomised, phase 2, open-label trial. Lancet. 2019 May 18;393(10185):2051-2058. doi: 10.1016/S0140-6736(18)32487-5. Epub 2019 Apr 11. PMID 30982687
- [Background] Iyengar P, All S, Berry MF, Boike TP, Bradfield L, Dingemans AC, Feldman J, Gomez DR, Hesketh PJ, Jabbour SK, Jeter M, Josipovic M, Lievens Y, McDonald F, Perez BA, Ricardi U, Ruffini E, De Ruysscher D, Saeed H, Schneider BJ, Senan S, Widder J, Guckenberger M. Treatment of Oligometastatic Non-Small Cell Lung Cancer: An ASTRO/ESTRO Clinical Practice Guideline. Pract Radiat Oncol. 2023 Sep-Oct;13(5):393-412. doi: 10.1016/j.prro.2023.04.004. Epub 2023 Apr 25. PMID 37294262
- [Background] Mitchell KG, Farooqi A, Ludmir EB, Corsini EM, Zhang J, Sepesi B, Vaporciyan AA, Swisher SG, Heymach JV, Zhang J, Gomez DR, Antonoff MB. Improved Overall Survival With Comprehensive Local Consolidative Therapy in Synchronous Oligometastatic Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2020 Jan;21(1):37-46.e7. doi: 10.1016/j.cllc.2019.07.007. Epub 2019 Aug 1. PMID 31447303
- [Background] Phillips R, Shi WY, Deek M, Radwan N, Lim SJ, Antonarakis ES, Rowe SP, Ross AE, Gorin MA, Deville C, Greco SC, Wang H, Denmeade SR, Paller CJ, Dipasquale S, DeWeese TL, Song DY, Wang H, Carducci MA, Pienta KJ, Pomper MG, Dicker AP, Eisenberger MA, Alizadeh AA, Diehn M, Tran PT. Outcomes of Observation vs Stereotactic Ablative Radiation for Oligometastatic Prostate Cancer: The ORIOLE Phase 2 Randomized Clinical Trial. JAMA Oncol. 2020 May 1;6(5):650-659. doi: 10.1001/jamaoncol.2020.0147. PMID 32215577
- [Background] Ruers T, Van Coevorden F, Punt CJ, Pierie JE, Borel-Rinkes I, Ledermann JA, Poston G, Bechstein W, Lentz MA, Mauer M, Folprecht G, Van Cutsem E, Ducreux M, Nordlinger B; European Organisation for Research and Treatment of Cancer (EORTC); Gastro-Intestinal Tract Cancer Group; Arbeitsgruppe Lebermetastasen und tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); National Cancer Research Institute Colorectal Clinical Study Group (NCRI CCSG). Local Treatment of Unresectable Colorectal Liver Metastases: Results of a Randomized Phase II Trial. J Natl Cancer Inst. 2017 Sep 1;109(9):djx015. doi: 10.1093/jnci/djx015. PMID 28376151
- [Background] Chmura S, Winter KA, Robinson C, Pisansky TM, Borges V, Al-Hallaq H, Matuszak M, Park SS, Yi S, Hasan Y, Bazan J, Wong P, Yoon HA, Horton J, Gan G, Milano MT, Sigurdson ER, Moughan J, Salama JK, White J. Evaluation of Safety of Stereotactic Body Radiotherapy for the Treatment of Patients With Multiple Metastases: Findings From the NRG-BR001 Phase 1 Trial. JAMA Oncol. 2021 Jun 1;7(6):845-852. doi: 10.1001/jamaoncol.2021.0687. PMID 33885704
- [Background] Luke JJ, Lemons JM, Karrison TG, Pitroda SP, Melotek JM, Zha Y, Al-Hallaq HA, Arina A, Khodarev NN, Janisch L, Chang P, Patel JD, Fleming GF, Moroney J, Sharma MR, White JR, Ratain MJ, Gajewski TF, Weichselbaum RR, Chmura SJ. Safety and Clinical Activity of Pembrolizumab and Multisite Stereotactic Body Radiotherapy in Patients With Advanced Solid Tumors. J Clin Oncol. 2018 Jun 1;36(16):1611-1618. doi: 10.1200/JCO.2017.76.2229. Epub 2018 Feb 13. PMID 29437535
- [Background] Onderdonk BE, Chmura SJ. The Yin and Yang of Cytoreductive SBRT in Oligometastases and Beyond. Front Oncol. 2019 Aug 2;9:706. doi: 10.3389/fonc.2019.00706. eCollection 2019. PMID 31428580
- [Background] Gustafson MP, Bornschlegl S, Park SS, Gastineau DA, Roberts LR, Dietz AB, Hallemeier CL. Comprehensive assessment of circulating immune cell populations in response to stereotactic body radiation therapy in patients with liver cancer. Adv Radiat Oncol. 2017 Aug 18;2(4):540-547. doi: 10.1016/j.adro.2017.08.003. eCollection 2017 Oct-Dec. PMID 29204520
- [Background] Ko EC, Raben D, Formenti SC. The Integration of Radiotherapy with Immunotherapy for the Treatment of Non-Small Cell Lung Cancer. Clin Cancer Res. 2018 Dec 1;24(23):5792-5806. doi: 10.1158/1078-0432.CCR-17-3620. Epub 2018 Jun 26. PMID 29945993
- [Background] Maehata Y, Onishi H, Kuriyama K, Aoki S, Araya M, Saito R, Tominaga L, Oguri M, Araki T. Immune responses following stereotactic body radiotherapy for stage I primary lung cancer. Biomed Res Int. 2013;2013:731346. doi: 10.1155/2013/731346. Epub 2013 Nov 10. PMID 24324972
- [Background] Wu L, Zhu J, Rudqvist NP, Welsh J, Lee P, Liao Z, Xu T, Jiang M, Zhu X, Pan X, Li P, Zhou Z, He X, Yin R, Feng J. T-Cell Receptor Profiling and Prognosis After Stereotactic Body Radiation Therapy For Stage I Non-Small-Cell Lung Cancer. Front Immunol. 2021 Oct 18;12:719285. doi: 10.3389/fimmu.2021.719285. eCollection 2021. PMID 34733273
- [Background] Luke JJ, Onderdonk BE, Bhave SR, Karrison T, Lemons JM, Chang P, Zha Y, Carll T, Krausz T, Huang L, Martinez C, Janisch LA, Hseu RD, Moroney JW, Patel JD, Khodarev NN, Salama JK, Ott PA, Fleming GF, Gajewski TF, Weichselbaum RR, Pitroda SP, Chmura SJ. Improved Survival Associated with Local Tumor Response Following Multisite Radiotherapy and Pembrolizumab: Secondary Analysis of a Phase I Trial. Clin Cancer Res. 2020 Dec 15;26(24):6437-6444. doi: 10.1158/1078-0432.CCR-20-1790. Epub 2020 Oct 7. PMID 33028595
- [Background] Bestvina CM, Pointer KB, Karrison T, Al-Hallaq H, Hoffman PC, Jelinek MJ, Juloori A, Melotek JM, Murgu S, Partouche J, Vokes EE, Weichselbaum RR, Pitroda SP, Patel JD, Chmura SJ. A Phase 1 Trial of Concurrent or Sequential Ipilimumab, Nivolumab, and Stereotactic Body Radiotherapy in Patients With Stage IV NSCLC Study. J Thorac Oncol. 2022 Jan;17(1):130-140. doi: 10.1016/j.jtho.2021.08.019. Epub 2021 Sep 6. PMID 34500113
- [Background] Yu J, Green MD, Li S, Sun Y, Journey SN, Choi JE, Rizvi SM, Qin A, Waninger JJ, Lang X, Chopra Z, El Naqa I, Zhou J, Bian Y, Jiang L, Tezel A, Skvarce J, Achar RK, Sitto M, Rosen BS, Su F, Narayanan SP, Cao X, Wei S, Szeliga W, Vatan L, Mayo C, Morgan MA, Schonewolf CA, Cuneo K, Kryczek I, Ma VT, Lao CD, Lawrence TS, Ramnath N, Wen F, Chinnaiyan AM, Cieslik M, Alva A, Zou W. Liver metastasis restrains immunotherapy efficacy via macrophage-mediated T cell elimination. Nat Med. 2021 Jan;27(1):152-164. doi: 10.1038/s41591-020-1131-x. Epub 2021 Jan 4. PMID 33398162
- [Background] Rokni MB, Pointer KB, George J, Luke JJ, Chmura SJ, Redler G. Radiation treatment planning study to investigate feasibility of delivering Immunotherapy in Combination with Ablative Radiosurgery to Ultra-High DoSes (ICARUS). J Appl Clin Med Phys. 2021 Mar;22(3):196-206. doi: 10.1002/acm2.13204. Epub 2021 Feb 24. PMID 33626240
- [Background] Bergsma DP, Salama JK, Singh DP, Chmura SJ, Milano MT. The evolving role of radiotherapy in treatment of oligometastatic NSCLC. Expert Rev Anticancer Ther. 2015;15(12):1459-71. doi: 10.1586/14737140.2015.1105745. Epub 2015 Nov 4. PMID 26536370
- [Background] Timmerman R, Paulus R, Galvin J, Michalski J, Straube W, Bradley J, Fakiris A, Bezjak A, Videtic G, Johnstone D, Fowler J, Gore E, Choy H. Stereotactic body radiation therapy for inoperable early stage lung cancer. JAMA. 2010 Mar 17;303(11):1070-6. doi: 10.1001/jama.2010.261. PMID 20233825
- [Background] Rusthoven KE, Kavanagh BD, Cardenes H, Stieber VW, Burri SH, Feigenberg SJ, Chidel MA, Pugh TJ, Franklin W, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for liver metastases. J Clin Oncol. 2009 Apr 1;27(10):1572-8. doi: 10.1200/JCO.2008.19.6329. Epub 2009 Mar 2. PMID 19255321
- [Background] Demaria S, Kawashima N, Yang AM, Devitt ML, Babb JS, Allison JP, Formenti SC. Immune-mediated inhibition of metastases after treatment with local radiation and CTLA-4 blockade in a mouse model of breast cancer. Clin Cancer Res. 2005 Jan 15;11(2 Pt 1):728-34. PMID 15701862
- [Background] Packard BZ, Toptygin DD, Komoriya A, Brand L. Profluorescent protease substrates: intramolecular dimers described by the exciton model. Proc Natl Acad Sci U S A. 1996 Oct 15;93(21):11640-5. doi: 10.1073/pnas.93.21.11640. PMID 8876189
- [Background] McBride WH, Chiang CS, Olson JL, Wang CC, Hong JH, Pajonk F, Dougherty GJ, Iwamoto KS, Pervan M, Liao YP. A sense of danger from radiation. Radiat Res. 2004 Jul;162(1):1-19. doi: 10.1667/rr3196. PMID 15222781
- [Background] Durante M, Reppingen N, Held KD. Immunologically augmented cancer treatment using modern radiotherapy. Trends Mol Med. 2013 Sep;19(9):565-82. doi: 10.1016/j.molmed.2013.05.007. Epub 2013 Jul 4. PMID 23831337
- [Background] Gaipl US, Multhoff G, Scheithauer H, Lauber K, Hehlgans S, Frey B, Rodel F. Kill and spread the word: stimulation of antitumor immune responses in the context of radiotherapy. Immunotherapy. 2014;6(5):597-610. doi: 10.2217/imt.14.38. PMID 24896628
- [Background] Demaria S, Formenti SC. Radiation as an immunological adjuvant: current evidence on dose and fractionation. Front Oncol. 2012 Oct 26;2:153. doi: 10.3389/fonc.2012.00153. eCollection 2012. PMID 23112958
- [Background] Akanda ZZ, Neeson PJ, John T, Barnett S, Hanna GG, Miller A, Jennens R, Siva S. A narrative review of combined stereotactic ablative radiotherapy and immunotherapy in metastatic non-small cell lung cancer. Transl Lung Cancer Res. 2021 Jun;10(6):2766-2778. doi: 10.21037/tlcr-20-1117. PMID 34295676
- [Background] Redmond KJ, Sahgal A, Foote M, Knisely J, Gerszten PC, Chao ST, Suh JH, Sloan AE, Chang EL, Machtay M, Lo SS. Single versus multiple session stereotactic body radiotherapy for spinal metastasis: the risk-benefit ratio. Future Oncol. 2015;11(17):2405-15. doi: 10.2217/fon.15.160. Epub 2015 Sep 15. PMID 26369361
- [Background] Hartsell WF, Scott CB, Bruner DW, Scarantino CW, Ivker RA, Roach M 3rd, Suh JH, Demas WF, Movsas B, Petersen IA, Konski AA, Cleeland CS, Janjan NA, DeSilvio M. Randomized trial of short- versus long-course radiotherapy for palliation of painful bone metastases. J Natl Cancer Inst. 2005 Jun 1;97(11):798-804. doi: 10.1093/jnci/dji139. PMID 15928300
- [Background] Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, Park K, Smith D, Artal-Cortes A, Lewanski C, Braiteh F, Waterkamp D, He P, Zou W, Chen DS, Yi J, Sandler A, Rittmeyer A; POPLAR Study Group. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1837-46. doi: 10.1016/S0140-6736(16)00587-0. Epub 2016 Mar 10. PMID 26970723
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Chen DS, Irving BA, Hodi FS. Molecular pathways: next-generation immunotherapy--inhibiting programmed death-ligand 1 and programmed death-1. Clin Cancer Res. 2012 Dec 15;18(24):6580-7. doi: 10.1158/1078-0432.CCR-12-1362. Epub 2012 Oct 19. PMID 23087408
- [Background] Blank C, Gajewski TF, Mackensen A. Interaction of PD-L1 on tumor cells with PD-1 on tumor-specific T cells as a mechanism of immune evasion: implications for tumor immunotherapy. Cancer Immunol Immunother. 2005 Apr;54(4):307-14. doi: 10.1007/s00262-004-0593-x. Epub 2004 Dec 15. PMID 15599732
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] Wang JH, Wu Q, Yang P, Li H, Li J, Mountz JD, Hsu HC. Type I interferon-dependent CD86(high) marginal zone precursor B cells are potent T cell costimulators in mice. Arthritis Rheum. 2011 Apr;63(4):1054-64. doi: 10.1002/art.30231. PMID 21225691
- [Background] Blank C, Mackensen A. Contribution of the PD-L1/PD-1 pathway to T-cell exhaustion: an update on implications for chronic infections and tumor evasion. Cancer Immunol Immunother. 2007 May;56(5):739-45. doi: 10.1007/s00262-006-0272-1. Epub 2006 Dec 29. PMID 17195077
- [Background] Sun R, Limkin EJ, Vakalopoulou M, Dercle L, Champiat S, Han SR, Verlingue L, Brandao D, Lancia A, Ammari S, Hollebecque A, Scoazec JY, Marabelle A, Massard C, Soria JC, Robert C, Paragios N, Deutsch E, Ferte C. A radiomics approach to assess tumour-infiltrating CD8 cells and response to anti-PD-1 or anti-PD-L1 immunotherapy: an imaging biomarker, retrospective multicohort study. Lancet Oncol. 2018 Sep;19(9):1180-1191. doi: 10.1016/S1470-2045(18)30413-3. Epub 2018 Aug 14. PMID 30120041
- [Background] Korpics MC, Polley MY, Bhave SR, Redler G, Pitroda SP, Luke JJ, Chmura SJ. A Validated T Cell Radiomics Score Is Associated With Clinical Outcomes Following Multisite SBRT and Pembrolizumab. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):189-195. doi: 10.1016/j.ijrobp.2020.06.026. Epub 2020 Jun 20. PMID 32569799
- [Background] Sun R, Sundahl N, Hecht M, Putz F, Lancia A, Rouyar A, Milic M, Carre A, Battistella E, Alvarez Andres E, Niyoteka S, Romano E, Louvel G, Durand-Labrunie J, Bockel S, Bahleda R, Robert C, Boutros C, Vakalopoulou M, Paragios N, Frey B, Soria JC, Massard C, Ferte C, Fietkau R, Ost P, Gaipl U, Deutsch E. Radiomics to predict outcomes and abscopal response of patients with cancer treated with immunotherapy combined with radiotherapy using a validated signature of CD8 cells. J Immunother Cancer. 2020 Nov;8(2):e001429. doi: 10.1136/jitc-2020-001429. PMID 33188037
- [Background] Nioche C, Orlhac F, Boughdad S, Reuze S, Goya-Outi J, Robert C, Pellot-Barakat C, Soussan M, Frouin F, Buvat I. LIFEx: A Freeware for Radiomic Feature Calculation in Multimodality Imaging to Accelerate Advances in the Characterization of Tumor Heterogeneity. Cancer Res. 2018 Aug 15;78(16):4786-4789. doi: 10.1158/0008-5472.CAN-18-0125. Epub 2018 Jun 29. PMID 29959149
- [Background] Tamminga M, de Wit S, Schuuring E, Timens W, Terstappen LWMM, Hiltermann TJN, Groen HJM. Circulating tumor cells in lung cancer are prognostic and predictive for worse tumor response in both targeted- and chemotherapy. Transl Lung Cancer Res. 2019 Dec;8(6):854-861. doi: 10.21037/tlcr.2019.11.06. PMID 32010564
- [Background] Morgan TM, Wang X, Qian X, Switchenko JM, Nie S, Patel KR, Cassidy RJ, Shin DM, Beitler JJ. Measurement of circulating tumor cells in squamous cell carcinoma of the head and neck and patient outcomes. Clin Transl Oncol. 2019 Mar;21(3):342-347. doi: 10.1007/s12094-018-1930-4. Epub 2018 Aug 6. PMID 30084036
- [Background] Yu M. Metastasis Stemming from Circulating Tumor Cell Clusters. Trends Cell Biol. 2019 Apr;29(4):275-276. doi: 10.1016/j.tcb.2019.02.001. Epub 2019 Feb 21. PMID 30799250
- [Background] Rodrigues P, Vanharanta S. Circulating Tumor Cells: Come Together, Right Now, Over Metastasis. Cancer Discov. 2019 Jan;9(1):22-24. doi: 10.1158/2159-8290.CD-18-1285. PMID 30626605
- [Background] Gan GN, Eagles J, Keysar SB, Wang G, Glogowska MJ, Altunbas C, Anderson RT, Le PN, Morton JJ, Frederick B, Raben D, Wang XJ, Jimeno A. Hedgehog signaling drives radioresistance and stroma-driven tumor repopulation in head and neck squamous cancers. Cancer Res. 2014 Dec 1;74(23):7024-36. doi: 10.1158/0008-5472.CAN-14-1346. Epub 2014 Oct 8. PMID 25297633
- [Background] Gan GN, Jimeno A. Emerging from their burrow: Hedgehog pathway inhibitors for cancer. Expert Opin Investig Drugs. 2016 Oct;25(10):1153-66. doi: 10.1080/13543784.2016.1216973. Epub 2016 Aug 5. PMID 27459882
- [Background] Mego M, Karaba M, Minarik G, Benca J, Silvia J, Sedlackova T, Manasova D, Kalavska K, Pindak D, Cristofanilli M, Reuben JM, Mardiak J. Circulating Tumor Cells With Epithelial-to-mesenchymal Transition Phenotypes Associated With Inferior Outcomes in Primary Breast Cancer. Anticancer Res. 2019 Apr;39(4):1829-1837. doi: 10.21873/anticanres.13290. PMID 30952723
- [Background] Oweida A, Lennon S, Calame D, Korpela S, Bhatia S, Sharma J, Graham C, Binder D, Serkova N, Raben D, Heasley L, Clambey E, Nemenoff R, Karam SD. Ionizing radiation sensitizes tumors to PD-L1 immune checkpoint blockade in orthotopic murine head and neck squamous cell carcinoma. Oncoimmunology. 2017 Aug 3;6(10):e1356153. doi: 10.1080/2162402X.2017.1356153. eCollection 2017. PMID 29123967
- [Background] Oweida A, Hararah MK, Phan A, Binder D, Bhatia S, Lennon S, Bukkapatnam S, Van Court B, Uyanga N, Darragh L, Kim HM, Raben D, Tan AC, Heasley L, Clambey E, Nemenoff R, Karam SD. Resistance to Radiotherapy and PD-L1 Blockade Is Mediated by TIM-3 Upregulation and Regulatory T-Cell Infiltration. Clin Cancer Res. 2018 Nov 1;24(21):5368-5380. doi: 10.1158/1078-0432.CCR-18-1038. Epub 2018 Jul 24. PMID 30042205
- [Background] Cheng Y, Wang T, Lv X, Li R, Yuan L, Shen J, Li Y, Yan T, Liu B, Wang L. Detection of PD-L1 Expression and Its Clinical Significance in Circulating Tumor Cells from Patients with Non-Small-Cell Lung Cancer. Cancer Manag Res. 2020 Mar 19;12:2069-2078. doi: 10.2147/CMAR.S245425. eCollection 2020. PMID 32256114
- [Background] Berggren KL, Restrepo Cruz S, Hixon MD, Cowan AT, Keysar SB, Craig S, James J, Barry M, Ozbun MA, Jimeno A, McCance DJ, Beswick EJ, Gan GN. MAPKAPK2 (MK2) inhibition mediates radiation-induced inflammatory cytokine production and tumor growth in head and neck squamous cell carcinoma. Oncogene. 2019 Nov;38(48):7329-7341. doi: 10.1038/s41388-019-0945-9. Epub 2019 Aug 15. PMID 31417185
- [Background] Witek MA, Aufforth RD, Wang H, Kamande JW, Jackson JM, Pullagurla SR, Hupert ML, Usary J, Wysham WZ, Hilliard D, Montgomery S, Bae-Jump V, Carey LA, Gehrig PA, Milowsky MI, Perou CM, Soper JT, Whang YE, Yeh JJ, Martin G, Soper SA. Discrete microfluidics for the isolation of circulating tumor cell subpopulations targeting fibroblast activation protein alpha and epithelial cell adhesion molecule. NPJ Precis Oncol. 2017;1:24. doi: 10.1038/s41698-017-0028-8. Epub 2017 Jul 25. PMID 29657983
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Rotz SJ, Leino D, Szabo S, Mangino JL, Turpin BK, Pressey JG. Severe cytokine release syndrome in a patient receiving PD-1-directed therapy. Pediatr Blood Cancer. 2017 Dec;64(12). doi: 10.1002/pbc.26642. Epub 2017 May 24. PMID 28544595
- [Background] Adashek ML, Feldman M. Cytokine Release Syndrome Resulting From Anti-Programmed Death-1 Antibody: Raising Awareness Among Community Oncologists. J Oncol Pract. 2019 Sep;15(9):502-504. doi: 10.1200/JOP.19.00160. Epub 2019 Jul 16. No abstract available. PMID 31310573
- [Background] Merad M, Martin JC. Pathological inflammation in patients with COVID-19: a key role for monocytes and macrophages. Nat Rev Immunol. 2020 Jun;20(6):355-362. doi: 10.1038/s41577-020-0331-4. Epub 2020 May 6. PMID 32376901
- [Background] Riegler LL, Jones GP, Lee DW. Current approaches in the grading and management of cytokine release syndrome after chimeric antigen receptor T-cell therapy. Ther Clin Risk Manag. 2019 Feb 28;15:323-335. doi: 10.2147/TCRM.S150524. eCollection 2019. PMID 30880998
- [Background] Ravelli A, Minoia F, Davi S, Horne A, Bovis F, Pistorio A, Arico M, Avcin T, Behrens EM, De Benedetti F, Filipovic L, Grom AA, Henter JI, Ilowite NT, Jordan MB, Khubchandani R, Kitoh T, Lehmberg K, Lovell DJ, Miettunen P, Nichols KE, Ozen S, Pachlopnik Schmid J, Ramanan AV, Russo R, Schneider R, Sterba G, Uziel Y, Wallace C, Wouters C, Wulffraat N, Demirkaya E, Brunner HI, Martini A, Ruperto N, Cron RQ; Paediatric Rheumatology International Trials Organisation; Childhood Arthritis and Rheumatology Research Alliance; Pediatric Rheumatology Collaborative Study Group; Histiocyte Society. 2016 Classification Criteria for Macrophage Activation Syndrome Complicating Systemic Juvenile Idiopathic Arthritis: A European League Against Rheumatism/American College of Rheumatology/Paediatric Rheumatology International Trials Organisation Collaborative Initiative. Ann Rheum Dis. 2016 Mar;75(3):481-9. doi: 10.1136/annrheumdis-2015-208982. PMID 26865703
- [Background] La Rosee P. Treatment of hemophagocytic lymphohistiocytosis in adults. Hematology Am Soc Hematol Educ Program. 2015;2015:190-6. doi: 10.1182/asheducation-2015.1.190. PMID 26637720
- [Background] Schram AM, Berliner N. How I treat hemophagocytic lymphohistiocytosis in the adult patient. Blood. 2015 May 7;125(19):2908-14. doi: 10.1182/blood-2015-01-551622. Epub 2015 Mar 10. PMID 25758828
- [Background] La Rosee P, Horne A, Hines M, von Bahr Greenwood T, Machowicz R, Berliner N, Birndt S, Gil-Herrera J, Girschikofsky M, Jordan MB, Kumar A, van Laar JAM, Lachmann G, Nichols KE, Ramanan AV, Wang Y, Wang Z, Janka G, Henter JI. Recommendations for the management of hemophagocytic lymphohistiocytosis in adults. Blood. 2019 Jun 6;133(23):2465-2477. doi: 10.1182/blood.2018894618. Epub 2019 Apr 16. PMID 30992265
- See also: National Institute of Health/National Cancer Institute - Cancer Therapy Evaluation Program (CTEP). Common Terminology Criteria for Adverse Events (CTCAE) — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_60
- See also: Study of PD1 Blockade by Pembrolizumab With Stereotactic Body Radiotherapy in Advanced Solid Tumors — https://clinicaltrials.gov/ct2/show/NCT02608385
- See also: Frebel H, Nindl V, Schuepbach RA, et al. Programmed death 1 protects from fatal circulatory failure during systemic virus infection of mice — https://pubmed.ncbi.nlm.nih.gov/23230000/
- See also: McClain KL, Eckstein O. Clinical features and diagnosis of hemophagocytic lymphohistiocytosis — https://www.uptodate.com/contents/clinical-features-and-diagnosis-of-hemophagocytic-lymphohistiocytosis